CLINICAL TRIAL: NCT02993848
Title: North American Scapula Consortium
Acronym: NASCon
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: North American Scapula Consortium (Other)
Collaborators: DePuy Synthes (Industry); Oregon Health and Science University (Other); University of Minnesota (Other)
Responsible Party: Principal Investigator, Peter A Cole, MD, Chair, Orthopaedic Dept., Regions Hospital; Professor, University of Minnesota, University of Minnesota
Other Study IDs: CON48716
Record Dates: First submitted 2016-12-05; First posted 2016-12-15 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Scapular Fracture
Keywords: Scapula; Fracture
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Operative Scapula Fracture: No intervention. Inclusion criteria and data collection is the same for both cohort.
  Interventions: Other: No intervention
- Non-Operative Scapula Fracture: No intervention. Inclusion criteria and data collection is the same for both cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The North American Scapula Consortium (NASCon) is a multi-center injury specific outcomes registry.

There currently exists a paucity of outcomes data in the literature on this patient population. The NASCon registry will be a resource in which investigators can conduct adequately powered clinical outcomes research resulting in higher quality research with meaningful results, improved patient care, and evidence-based advancement for the treatment of scapula fractures. Registries can lead to significant discoveries in comparative effectiveness specifically in areas where randomized control studies are not possible. Collecting post-treatment (operative and non-operative) patient outcome data for similar injury patterns has been shown effective in uncovering optimal standards for treatment.

DETAILED DESCRIPTION:
Number of Subjects:

Estimated

Year 1 10 Sites 80 Subjects Enrolled

Year 2 13 Sites 130 Subjects Enrolled

Year 3 16 Sites 170 Subjects Enrolled

Year 4 and on going 200 Subjects per year

The North American Scapula Consortium, NASCon is a multi center injury specific outcomes registry. Patients presenting to participating surgeons with Extra Articular and/or Intra Articular scapula fracture meeting inclusion criteria will be asked for their signed consent to participate in the outcomes registry regardless of treatment plan (operative or non-operative).

Justification for stated number of subjects:

The goal of this study is to capture as many patients meeting inclusion criteria from the enrolling sites as possible. The investigators estimate this to be between 10 and 13 patients per site, per year.

Participating sites: Participating sites will be identified based on their experience and expertise in scapula repair, their interest in research, and their desire to advance knowledge and continuing education in this area. Initially, Dr. Peter Cole will personally invite new sites. Future site recruitment will be approved by Dr. Peter Cole and a selected board. Sites must have the necessary research infrastructure and be willing and able to follow all rules and regulations associated with Human Research requirements. They will be required to submit evidence of site IRB approval prior to initiation.

Data Collection:

Time point: Day 0

Activity: obtain patient consent, x-rays, chart review, data pull from electronic medical record

Activity conducted by: study coordinator at participating NASCon site

Time point: 6 wks , 3 mos, 6 mos, 12 mos, 24 mos

Activity: patient questionnaires, Range of Motion, Strength, and x-rays

The following is a list of demographic and treatment variables that will be collected during the patient's initial enrollment visit as well as from the patient's EMR:

Demographics: Gender, date of birth, dominant hand

Injury: Inclusion indication, radiographic image, date of injury, mechanism of injury, side of scapular injury, ipsilateral UE fractures, other SSSC lesions, other system injuries, Ada & AO/OTA Classifications, prior treatment, and workman's compensation status.

Surgical Data (when applicable): Date of surgery, operative time, estimated blood loss, other procedures, subsequent shoulder procedures required, scapula operative approach, type of implant.

The following is a list of outcome variables that will be collected during each follow-up clinic visit as well as from the patient's EMR:

General Information: Physical Therapy, activity level, return to work, pain/pain medication, complications, subsequent procedures, radiographic image.

Range of Motion:

A 14 inch goniometer will be used to evaluate flexion, abduction, external rotation, internal rotation on injured and contralateral shoulder.

Strength:

A handheld dynamometer (MicroFET 2, Hoggan Health Industries, Draper, Utah), which has been previously published as a reliable technique10, will assess strength in shoulder flexion, abduction, and external rotation on injured and contralateral shoulder.

Disabilities of the Arm, Shoulder, and Hand questionnaire (DASH). 11

The DASH was developed to measure physical disability and symptoms of the upper extremities in people with upper extremity disorders (hand, wrist, elbow, and shoulder). It is a 30-item scale that addresses difficulty in performing various physical activities that require upper extremity function, stiffness, and impact of disability and symptoms on social activities, work, sleep, and psychological well-being. The score ranges from 0 to 100, where 0 is equivalent to no disability and 100 is equivalent to most severe disability. The DASH is a validated instrument with established normative and minimal clinically important difference.

SF-12v2

The SF-12v2 is a multipurpose, short-form health survey with 12 questions. The SF-12v2 was developed in 1994 by The Health Institute as a shortened version of the SF-36 health survey. It yields an eight-scale profile of scores as well as physical and mental health summary measures. The eight scales include: physical functioning, role of physical functioning, mental functioning, role of mental functioning, social function, bodily pain, vitality, and general health. It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group.

Reporting of Results:

Demographic data, treatment details, and outcome variables will be summarized through frequencies and proportions, if they are categorical, or through measures of central tendency (e.g., mean, median) and dispersion (e.g. standard deviation, quartiles) if they are continuous. Quarterly registry reporting will include enrollment rates, follow-up capture rates, descriptive summaries of demographic, surgical and outcomes data as well as a description of any safety events for which the membership or the sponsors should be made aware. Reports will be shared with the membership and study sponsors on a minimum of an annual basis.

Publication and presentation of outcomes is expected in peer-reviewed orthopaedic journals and symposia, once substantial data collection and outcomes of ≥1 year post-injury are accomplished. Additionally, opportunities to describe the establishment of an injury specific consortium and registry, including experience, process and tools utilized in the development of such a registry, may be pursued by the membership.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 yrs of age
* Operative and non-operative fractures meeting any one of the following criteria:

  * Extra - Articular fracture indication (one or more of the following): Glenopolar angle <30°, Medialization >1cm, and Angulation >30°
  * Intra-Articular fracture indication: >2mm
  * Patient signed consent

Exclusion Criteria:

* Patients meeting operative criteria that are not able to understand the consent for research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The NASCon registry will include all qualifying, consented scapula fracture patients who present to the participating site PI's clinics or practices for treatment of a scapula fracture. All site PIs will use the same standardized measurement tools (Glenopolar angle, Medialization, and Angulation) to evaluate participants.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Data Submission measured by total number of participating sites and patient enrollment | Three years
  Anticipated:
  Year 1 - 10 Sites,80 Subjects Enrolled Year 2 - 13 Sites, 130 Subjects Enrolled Year 3 - 16 Sites, 170 Subjects Enrolled

SECONDARY OUTCOMES:
Optimization of data submission and data collected by statistician review of exported data collection | Biannual review (June 2017, Dec 2017, June 2018, Dec 2018, June 2019, Dec 2019-end date)
  A qualified statistician will review all data submitted biannually and determine the percent of unpopulated fields and provide strategy for optimizing data collection. Sites will be notified of missing data and strongly encourages to complete.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Cole, MD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No